CLINICAL TRIAL: NCT05532384
Title: Effect of Early Postoperative Drinking Water on Postoperative Recovery Quality of Patients With Thyroid Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ZS-3566
Record Dates: First submitted 2022-08-30; First posted 2022-09-08 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-06

CONDITIONS: Thyroid Tumor
Keywords: Thyroidectomy; Enhanced Recovery After Surgery; Quality of Recovery-15
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial：Participants who enroll in RCTs differ from one another in known and unknown ways that can influence study outcomes, and yet cannot be directly controlled. By randomly allocating participants among compared treatments, an RCT enables statistical control over these influences. Provided it is designed well, conducted properly, and enrolls enough participants, an RCT may achieve sufficient control over these confounding factors to deliver a useful comparison of the treatments studied.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The anesthesiologists will obtain the group of patients through computer randomization before the patients leave the Post-Anesthesia Care Unit, and guide the patients to drink water. The questionnaire collectors and outcomes assessor will not be informed of the group of patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early resumption of oral intake (Experimental): Drink 30-50ML of normal temperature water after meeting the PACU transfer out standard. If the patient swallows successfully and does not cough, after returning to the ward, the medical staff of the ward will guide him or her to resume drinking and eating early: patient will resume drinking water within one hour after returning to the ward, a small amount of water for many times until the amount of drinking water reaches 300ml. If the patient does not have discomfort symptoms, he or she will resume eating according to normal drinking and eating habits.
  Interventions: Behavioral: Early resumption of oral intake
- Late resumption of oral intake (Other): Drink 30-50ML of normal temperature water after 6h after the operation. A small amount of water can be used several times, and the amount of water can reach 300ml. If the patient does not have any discomfort symptoms, it can guide the patient to recover diet according to his/her normal eating habits.
  Interventions: Behavioral: Late resumption of oral intake

INTERVENTIONS:
Behavioral: Early resumption of oral intake — as above
  Arms: Early resumption of oral intake
Behavioral: Late resumption of oral intake — as above
  Arms: Late resumption of oral intake

SUMMARY:
This study is a single-center, prospective and randomized controlled study to investigate the effects of early recovery of oral intake (E) and late recovery of oral intake (L) on postoperative recovery quality and satisfaction of patients undergoing thyroid surgery. The study's primary outcome is quality of recovery-15 scale (Qor-15).

DETAILED DESCRIPTION:
The subjects of this study are patients who will receive thyroid surgery in Peking Union Medical College Hospital. After the patient is included in the experiment, when the patient meets the exit criteria of the PACU, the patient will be randomly assigned to early resumption of oral intake group and late resumption of oral intake group to receive different treatments. Finally, researchers will collecte and evaluate the different outcome indicators of the two groups of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. ASA Physical Status I-II
3. Body mass index 18.5-29.9kg/m2
4. First operation on operation day
5. Thyroid surgery

Exclusion Criteria:

1. Patients or family members cannot understand the conditions and objectives of this study
2. Preoperative patients with acute pharyngitis, hoarseness, cough, dysphagia, and high risk of aspiration
3. The surgeons or anesthesiologists point out that the patient is not suitable for early postoperative drinking (such as considering the injury of recurrent laryngeal nerve or lymphatic vessels during the operation)
4. Exclusion criteria of QoR-15* (*QoR-15 exclusion criteria: 1. Unable to understand words and language; 2. Difficult to cooperate due to mental disorders; 3. History of alcohol or drug abuse; 4. Any serious pre-existing medical condition that can limit the objective evaluation after surgery; 5. Any life-threatening complications; 6. Emergency surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
QoR-15 score on the first day after surgery | one day
  Using QoR-15 questionnaire to evaluate the quality of perioperative recovery. QoR-15 consists of 15 comprehensive questions, including physical comfort (5 items), psychological support (2 items), physical independence (2 items), emotional state (4 items), and pain (2 items), each item is scored with 0-10 points, 0 represents poor state, 10 represents good state, and the total score is the QoR-15 score of the patient.

SECONDARY OUTCOMES:
QoR-15 score on the day of discharge | one day
  Using QoR-15 questionnaire to evaluate the quality of perioperative recovery. QoR-15 consists of 15 comprehensive questions, including physical comfort (5 items), psychological support (2 items), physical independence (2 items), emotional state (4 items), and pain (2 items), each item is scored with 0-10 points, 0 represents poor state, 10 represents good state, and the total score is the QoR-15 score of the patient.
Patient satisfaction | through patient discharge, an average of 3-4 day
  The overall satisfaction of the patients during hospitalization was scored immediately before the patients were discharged from the hospital. The patients were scored according to 0-10 points, 0 being completely dissatisfied and 10 being completely satisfied.
Postoperative pain | through patient discharge, an average of 3-4 day
  The patients were given self-evaluation before the first drinking water and 8 hours after the operation. They were divided into pharyngeal pain and surgical incision pain, which were scored according to 0-10 points respectively. 0 point was completely painless, and 10 point was unbearable pain.
Recovery of digestive function | through recovery of digestive function, an average of 1-2 day after surgery
  Postoperative defecation and exhaustion time
Length of hospital stay | through patient discharge, an average of 3-4 day
  Length of hospital stay
Total drainage volume after operation | through removal of drainage tube, an average of 2 day
  Total drainage volume after operation

CONTACTS AND LOCATIONS:
Overall Officials: Shen Le, PhD, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Wu Juelun, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No